CLINICAL TRIAL: NCT02746549
Title: Randomized, Clinical Study to Compare Accuracy of 1.5 T Versus 3 T Magnetic Resonance Arterial Spin Labeling to Measure Renal Blood Flow and the Changes of Renal Perfusion Caused by Physiological Stress (Cold Pressor Test).
Brief Title: Accuracy of 1.5 T Versus 3 T Magnetic Resonance Arterial Spin Labeling to Measure Renal Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MRT2014
Record Dates: First submitted 2015-10-08; First posted 2016-04-21 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Hypertension; Chronic Kidney Disease
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.5 Tesla MRI (Experimental): Measurement of renal perfusion by 1.5 Tesla MRI with arterial spin labelling
  Interventions: Other: renal perfusion
- 3.0 Tesla MRI (Experimental): Measurement of renal perfusion by 3.0 Tesla MRI with arterial spin labelling
  Interventions: Other: renal perfusion

INTERVENTIONS:
Other: renal perfusion — measurement of renal perfusion with MRI arterial spin labelling technique

SUMMARY:
In this study we want to compare the accuracy of two methods to measure renal perfusion by MRI spin labelling technique: the first measurement done with the 1.5 T MRI versus the second one obtained with the 3.0 T MRI (Siemens MRI device).

Additionally we want to compare the changes of renal perfusion caused by physiological stress. The used stress test is the cold pressor test done at the forehead.

DETAILED DESCRIPTION:
Magnetic resonance imaging based arterial spin labeling is a technique to measure renal blood flow. Renal perfusion measurement is an important tool to analyze renal function and to detect acute kidney injury. The perfusion measurement is based on two data acquisitions, one with a global inversion prepulse followed by one with a slice selective prepulse (FAIR). The prepulses lead to a labeling of blood water spins. In contrast to the global inversion prepulse, the slice selective inversion prepulse only labels the blood water spins inside the kidney but not the inflowing blood water spins. Subtraction of both images therefore reflects the local perfusion. A third image without the FAIR preparation pulse is measured to normalize the signal intensifiers on each patients.

MRI based arterial spin labeling is a noninvasive assessment not using contrast agents to measure the functional parameters of the kidney. This is avoiding serious complications such as acute kidney failure and nephrogenic systemic fibrosis. There is no known negative impact to the patient. In addition we now want to analyze the validity of this MRI-technique by provoking acutely changes of renal plasma flow. As a further provocative maneuver we selected the cold pressor test as a physiological stress test. Forehead cooling activates the sympathetic nervous system and increases blood pressure and heart rate by causing pain. This mechanism has got an impact on renal haemodynamics. To minimize the possible cold injuries we use the 1°C ice water pack only for 60 seconds and avoid the contact to the eyes.

In this study we want to compare the accuracy of two methods to measure renal perfusion by MRI spin labelling technique: the first measurement done with the 1.5 T MRI versus the second one obtained with the 3.0 T MRI (Siemens MRI device).

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients are eligible. Females of child bearing potential (WOCBP) are only eligible if pregnancy test at the screening visit is negative and they use adequate contraceptive precautions during the trial.
* Healthy volunteers and patients who have hypertension stage 1 or 2 or patients who have diabetes at a max of 2 oral antidiabetic agents will be included

Exclusion Criteria:

* eGFR ≤ 45 ml/min/1.75m²
* any cardiovascular or cerebrovascular other other severe events within the last 3 months
* arterial hypertension grad > 2 ( blood pressure ≥ 180/110)
* Subject who do not give written consent, that pseudonymous data will be transferred in line with the duty of documentation and the duty of notification according to § 12 and § 13 GCP-V
* Any contraindications to MRI
* Brain aneurysm clip
* Implanted cardiac pacemaker, pacemaker wires or defibrillator
* Prosthetic heart valves
* Cochlear implant
* Ocular foreign body
* Implanted insulin pump,
* Tattoo (as determined by imager)
* agoraphobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of 1.5 T versus 3 T magnetic resonance arterial spin labeling to measure renal perfusion (ml/min) | 2 weeks
  Renal function will be measured in ml/min by MRI arterial spin labelling technique.

CONTACTS AND LOCATIONS:
Overall Officials: Roland E. Schmieder, MD, Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- Clinical Research Unit, Department of Nephrology and Hypertension, University of Erlangen-Nürnberg, Erlangen, Germany

REFERENCES:
- [Background] Hammon M, Janka R, Siegl C, Seuss H, Grosso R, Martirosian P, Schmieder RE, Uder M, Kistner I. Reproducibility of Kidney Perfusion Measurements With Arterial Spin Labeling at 1.5 Tesla MRI Combined With Semiautomatic Segmentation for Differential Cortical and Medullary Assessment. Medicine (Baltimore). 2016 Mar;95(11):e3083. doi: 10.1097/MD.0000000000003083. PMID 26986143